CLINICAL TRIAL: NCT00297635
Title: Telemetric Glucose Data Acquisition During Initiation of Insulin Pump Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Decided not to participate in study per Leslie Padron-Massaro
Sponsor: Thomas Jefferson University (Other)
Collaborators: LifeScan (Industry); Diabetech (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06C.07
Record Dates: First submitted 2006-02-23; First posted 2006-02-28 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Insulin-Dependent
Keywords: Hyperglycemia; Insulin Infusion Systems; Blood Glucose Self-Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia

INTERVENTIONS:
Device: GlucoDYNAMIX™ intervention system
Device: GlucoMON™ telemetry device

SUMMARY:
This study will help determine whether the use of a wireless glucose meter and and an internet-based automated diabetes management system to organize blood glucose values will help improve glucose control during the start of continuous subcutaneous insulin infusion therapy by an insulin pump device in patients with type 1 diabetes. Outcome measures to be determined include an assessment of glucose excursions, overall glucose control, health care team staff and patient time required and a satisfaction survey.

DETAILED DESCRIPTION:
The study is focused on the following objectives:

1. Determine whether the use of the GlucoDYNAMIX™ diabetes intervention system and the GlucoMON™ telemetry device will facilitate faster regulation of blood glucose excursions into a well-controlled range, compared to conventional monitoring and reporting.

   * hemoglobin A1c at the end of the 3 month study period and again after an additional 3 month follow-up period to account for a possible for an extended difference between the groups;
   * magnitude of glucose excursions and fluctuations as indicated by the standard deviation between glucose tests to indicate relative glucose control and the mean daily glucose value over the 3 month period following the initiation of pump therapy; and,
   * frequency of severe hypoglycemia and extended hyperglycemia.
2. Determine whether use of the GlucoDYNAMIX intervention system, during initiation of adult insulin pump starts, results in a measured saving of staff time in support of data collection, analysis and patient feedback including delivery and follow-up to monitor effects on glucose control from patient implementation of prescribed changes. This objective will be measured by:

   * tracking the number of interventions each day;
   * estimating the amount of time spent collecting, analyzing and communicating with each study patient; and,
   * daily logs will be tallied and verified weekly.
3. To determine through use of questionnaires administered to the patients and to the professional staff whether use of the technology results in perceived improvement in the quality of care and improved satisfaction for all involved. This objective is primarily concerned with people's willingness to commit to using a similar technology as standard practice for future initiation of insulin pump starts for adult patient with diabetes mellitus.

Study Design and Description The study is designed to run for a period of 3 months of intensive management for each enrolled patient as they begin insulin pump therapy plus detailed glucose records beginning 4 weeks prior to the initiation of insulin pump therapy. Understanding relative glucose control following intensive management requires that we consider the results of the patient's HbA1c 3 months after conclusion of intensive management thus extending the time frame to 6 months.

Group A The Intervention Technology Group will be issued a GlucoMON device, a GlucoMON wall-mount recharging unit, a OneTouch Ultra glucose meter, paper logbook forms and test strips to support frequent testing for the 3 months following initiation of insulin pump therapy. The patient will be instructed on use and care of the GlucoMON as well as the OneTouch Ultra during a one-on-one session at the meeting immediately prior to initial delivery of insulin via the pump start.

Patients are also issued a specially configured low-cost 2way wireless email device which supports sending and receiving individual messages of up to 500 characters including the ability to send canned response options for easy data marking. Real-time messaging as part of the system is described in Addendum B. The intelligent logic behind the patient interaction is managed on a server in Diabetech's remote data center thus allowing for easy modification and centralized management of the patient interaction.

The TJU diabetes staff will initially review the patient record daily and will document the results of their review including any changes prescribed to the patient and the approximate amount of time involved in the handling of the encounter.

Group B (Control) The Conventional Technology Group will be issued a OneTouch Ultra glucose meter, paper logbook forms and test strips to support frequent testing for the 3 months following initiation of insulin pump therapy. The patient will be instructed on use and care of the OneTouch Ultra during a one-on-one session at the meeting to begin initial delivery of insulin via the pump start.

Patients will be instructed to complete the logbooks and fax daily to the TJU diabetes center. The TJU diabetes staff are available to review patient logs Monday thru Friday 8-5. Emergency after hours help is also available. The staff will initially review the patient logbook and will document the results of their review including any changes prescribed to the patient and the approximate amount of time involved in the handling of the encounter.

Data Analysis The data collected will include the patient's self-monitoring blood glucose (SMBG) test data, time-event logging annotations to the glucose tests, baseline and follow-up hemoglobin A1c test results, clinical events including hypoglycemia and hyperglycemia, and results of satisfaction questionnaires and time spent for analysis by the clinical staff for each patient.

The endpoints to be measured include frequent blood glucose testing, as is usual when a patient is initiating therapy with an insulin infusion pump, as well as HbA1c. The glucose levels will be analyzed with regard to the magnitude of glucose excursions and fluctuations and the mean daily glucose value over the 6 month period following the initiation of pump therapy.

The mean and standard deviation of each treatment group's (intervention and control) HbA1c will be calculated for each time point (0, 3, and 6 months post enrollment). Statistical differences in the HbA1c values between treatment groups at each time point and between different time points for each group will be sought. In addition, the change in HbA1c between time points (0 to 3, 3 to 6, and 0 to 6) will be calculated. The mean and standard deviation of these HbA1c changes will be calculated for each treatment group and analyzed for statistical significance.

SMBG data will be analyzed using glycemic control indices to compare the efficacy of both treatments. The following numerical indices will be used to describe the quality of metabolic control:

1. The mean and standard deviation of patient SMBG data
2. The percentage of SMBG data points that are above and below a threshold for hyperglycemia (e.g., 200mg/dl) and hypoglycemia (e.g., 60mg/dl)
3. The M-value is a quantitative index of the lack of treatment efficacy of an individual patient. The index describes both mean glycemic control and glucose excursions. The M-value is a logarithmic transformation of the deviation from an arbitrary standard (selected by the physician) that gives extra weight to hypoglycemic values. The original concept of Schlichtkrull et al. (1965)3 has been modified by Service et al. (1970) 4 into the formula:

   |10 log10 (x/standard)|3 / n where x is a SMBG data point, standard is aM = glucose value chosen to define the degree of metabolic control (typically 100 mg/dl), and n is the number of samples. BG values below 100mg/dl cause the M-value to rise rapidly while BG values above 100 mg/dl cause the M-value to rise more slowly. M-values less than 18 correspond to good metabolic control [Schlichtkrull J 1965].
4. The mean amplitude of glycemic excursions (MAGE) quantifies the amplitude and duration of wide swings of BG values, diurnal variability of mean BG values, and episodes of hypoglycemia as an index of diabetic instability. MAGE is calculated by taking the arithmetic mean of the changes in BG when they exceed one standard deviation of the BG mean over the preceding 24-hour period. Excursions less than 1 standard deviation are ignored. MAGE is a valuable index of metabolic control in healthy and diabetic subjects [Service 1970]. MAGE averaged 42 mg/dl in healthy subjects, 147 mg/dl in type 1 diabetic patients treated with multiple injections of short-acting insulin, and 161 mg/dl in type 1 diabetic patients treated with a single daily injection of intermediate-acting insulin.

These indices will be computed using a moving window of data. The window will be stepped across each patient's SMBG data set through the intensive management period. Those data points that fall within the window will be used to compute the indices. The steps and widths of the window will be set at 1, 7, 14, and 28 days. For example, with a step and width of 7 days, each calculation of the M-value of a patient's SMBG data would encompass 7 days and there would be 12 different calculations for each week of the 3-month intensive management period. Statistical differences in the indices for a given window for each treatment group will be sought.

The amount of time taken by nurses and physicians to manage each patient will be tabulated. These data will be used to compute a cost associated with the management of the insulin pump start for each patient. The mean and standard deviation of this cost will be calculated for each treatment group and analyzed for a statistical significance.

A paired Student t-test or a one-way analysis of variance will be used to calculate a significant difference. A p value less than 0.05 will be considered statistically significant.

Standard Care Guidelines typically involve the diabetes center distributing a handbook of sorts to the patient upon diagnosis or as part of the initial visit to your center. In terms of ongoing care, patients are responsible for acquiring tools on their own for managing diabetes. In addition to insulin, patients must purchase their own glucose meters, test strips, lancing device, lancets, alcohol, fast acting sugar of some sort to treat low blood sugar, glucagon for severe hypoglycemia, etc... Depending on the form of insulin therapy, the patient must also purchase syringes or an insulin pump with disposable cartridges and infusion sets.

For the duration of the study, patients enrolled as Standard Care (Group B) will be given a glucose meter and test strips at no charge.

To facilitate communication of blood sugars and other diabetes relevant data with the center, the diabetes center shares one page of a standardized logbook form on 8.5" x 11" paper. It is the patient's responsibility to make copies of this form for their own use and also to deliver these completed forms to the diabetes center as needed. Methods for delivering this logbook include faxing (a patient must purchase their own fax machine or pay/borrow as well as any costs associated with fax transmission), US Mail (using their own envelope and postage) or hand deliver (using their own transportation).

Study Population As a patient elects to participate they will be assigned alternatively to either Group A or Group B beginning with assignment of the first patient enrolled into Group A.

Informed Consent Informed consent will be obtained from each participant.

Documentation Requirements All data and documentation will be held private and secure in compliance with HIPAA guidelines.

References

1. Wireless Diabetes Management System; Poster Presentation 2003 Diabetes Technology Society: December 2002 - April 2003; Stephen Ponder MD CDE, Driscoll Children's Hospital with support from Diabetech.
2. Wojcicki JM, Analysis: Transfer of the Data Collected by the Patient to the Health Care Providers: Problems and Solutions, Diabetes Technology & Therapeutics. Apr 2005, Vol. 7, No. 2: 248-252
3. Schlichtkrull J. Munck O. Jersild M. The M-value, an index of blood-sugar control in diabetics. Acto Med Scand. 177(1):95-102, 1965.
4. Service FJ. Molnar GD. Rosevear JW. Ackerman E. Gatewood LC. Taylor WF. Mean amplitude of glycemic excursions, a measure of diabetic instability. Diabetes. 19(9):644-55, 1970

ELIGIBILITY:
Inclusion Criteria:

Patients must reside in the Philadelphia area and participate in regular in person visits to the Jefferson Diabetes Research Center. Patients must be at the stage of their treatment where they are going to initiate insulin infusion pump therapy. Patients must be at least 18 years of age before starting the protocol and must have never used an insulin pump before. Ideally, at least a few of the study participants will use English as a second language. Since the technology is capable of delivering messages to the wireless email device in several languages including Spanish and French, there is no English only requirement. Likewise, patients not capable of operating the wireless email device will be included since the GlucoMON device is specially designed to enable patient use without technology aptitude typical for personal computers and interactive wireless devices.

Exclusion Criteria:

Patients living outside the Philadelphia area and those that are not immediately going to initiate insulin pump therapy wil be excluded. Patients unwilling to perform at least 4 blood glucose self-tests will be ineligible for participation in this study. Conventional guidelines for minimum self-care will apply including criteria for discontinuance of insulin pump therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Regulation of blood glucose excursions, measured by hemoglobin A1c at the end of the 3 month study period and again after an additional 3 month follow-up period
Magnitude of glucose excursions and fluctuations as indicated by the standard deviation between glucose tests to indicate relative glucose control and the mean daily glucose value over the 3 month period following the initiation of pump therapy

SECONDARY OUTCOMES:
Frequency of severe hypoglycemia and extended hyperglycemia.
Saving of staff time in support of data collection, analysis and patient feedback including delivery and follow-up to monitor effects on glucose control from patient implementation of prescribed changes.
Whether use of the technology results in perceived improvement in the quality of care and improved satisfaction for all involved

CONTACTS AND LOCATIONS:
Overall Officials: Barry J. Goldstein, MD, PhD, Principal Investigator — Thomas Jefferson University

REFERENCES:
- See also: TJU Division of Endocrinology, Diabetes and Metabolic Diseases — http://www.jeffersonhospital.org/departments-and-services/diabetes-research-program.aspx
- See also: TJU Diabetes Research Center — http://www.jeffersonhospital.org/endocrinology/article4158.html